CLINICAL TRIAL: NCT01625260
Title: A Phase Ib/II Study of ALT-801 in Patients With Bacillus Calmette-Guerin (BCG) Failure Non-muscle Invasive Bladder Cancer
Brief Title: A Study of ALT-801 in Patients With Bacillus Calmette-Guerin (BCG) Failure Non-Muscle Invasive Bladder Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to low enrollment.
Sponsor: Altor BioScience (Industry)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-801-01-12
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: cancer; immunotherapy; targeted; non-muscle invasive; interleukin-2; antitumor; TCR; T-cell receptor; p53; p53 gene; p53 tumor supressor protein; urothelial cancer; bladder cancer; HLA-A2 positive; HLA-A*0201/p53 aa264-272; HLA complex; refractory; relapsed; BCG; multi-focal; carcinoma in situ; transitional cell carcinoma; gemcitabine
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Neoplasms; Urinary Bladder Neoplasms; Recurrence; Carcinoma in Situ; Carcinoma, Transitional Cell | interventions — ALT-801; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.06 mg/kg ALT-801 with 1000 mg/m^2 Gemcitabine (Experimental): ALT-801 at 0.06 mg/kg with Gemcitabine at 1000 mg/m^2
  Interventions: Biological: ALT-801; Drug: Gemcitabine
- 0.08 mg/kg ALT-801 with 1000 mg/m^2 Gemcitabine (Experimental): ALT-801 at 0.08 mg/kg with Gemcitabine at 1000 mg/m^2
  Interventions: Biological: ALT-801; Drug: Gemcitabine

INTERVENTIONS:
Biological: ALT-801 — Intravenous infusion: 2 treatment courses and 1 maintenance course; on Day 3, 5, 8 and 15 of each course.
  Other Names: c264scTCR-IL2
Drug: Gemcitabine — Intravenous infusion: 2 treatment courses and 1 maintenance course; on Day 1 and 8 of each course.

SUMMARY:
This is a Phase Ib/II, open-label, multi-center and competitive enrollment study of ALT-801 combined with gemcitabine for patients who have BCG failure (defined as refractory, relapsing or intolerant), non-muscle invasive bladder cancer and refuse or are not medically fit to undergo a radical cystectomy recommended by the participating urologist as the standard next therapy per urologic guidelines. The purpose of this study is to confirm the safety and tolerability of a well-tolerated dose level of ALT-801, to determine the Recommended Dose level (RD) and characterize the immunogenicity of ALT-801 combined with gemcitabine in treated patients. The anti-tumor responses will also be assessed.

DETAILED DESCRIPTION:
Bladder cancer is the fifth most common cancer in the United States with an estimated 71,000 new cases and approximately 14,000 deaths in 2009. Bladder cancer is also the costliest to treat per patient of all cancers, with annual direct medical expenditures in excess of $3.7 billion in the United States. This is largely because approximately 70% of all new cases of bladder cancer present as non-muscle invasive bladder cancer (NMIBC), which tends to recur, requiring repeated interventions and long-term follow-up.

Altor Bioscience Corp. has developed a tumor-targeted IL-2 fusion protein, ALT-801, comprising human recombinant IL-2 genetically linked to a TCR domain capable of binding a tumor associated human p53 peptide presented in the context of HLA-A2.

ALT-801 will be evaluated as to whether it can prevent disease progression and allow for bladder preservation to maintain the quality of life for patients with BCG failure, defined as refractory, relapsing or intolerant, non-muscle invasive bladder cancer who refuse or are not medically fit to undergo a radical cystectomy recommended by the participating urologist as the standard next therapy per urologic guidelines.

ELIGIBILITY:
ENTRY CRITERIA:

DISEASE CHARATERISTICS:

* Histologically confirmed high-risk (high grade Ta, T1 or carcinoma in situ, tumor >4 cm or multi-focal) transitional cell carcinoma s/p TURBT with no remaining resectable disease within 4 weeks of study entry
* Intolerant of treatment with BCG or failure (refractory or relapsing) of at least one prior treatment with BCG
* Refuse or intolerant of a radical cystectomy
* No Evidence of regional and/or distant metastasis

PRIOR/CONCURRENT THERAPY:

* No concurrent radiotherapy, other chemotherapy, or other immunotherapy
* No scheduled radiotherapy, chemotherapy, other immunotherapy, or surgery before the scheduled response evaluation
* Must have recovered from side effects of prior treatments
* No concurrent use of other investigational agents

PATIENT CHARACTERISTICS:

Age

• ≥ 18 years

Performance Status

• ECOG 0, 1, or 2

Bone Marrow Reserve

* Absolute neutrophil count (AGC/ANC) ≥ 1,000/uL
* Platelets ≥ 100,000/uL
* Hemoglobin ≥ 8 g/dL

Renal Function

• Glomerular Filtration Rate (GFR) ≥ 50mL/min

Hepatic Function

* Total bilirubin ≤ 2.0 X ULN
* AST, ALT, ALP ≤ 3.0 X ULN

Cardiovascular

* No congestive heart failure < 6 months
* No severe/unstable angina pectoris < 6 months
* No myocardial infarction < 6 months
* No history of ventricular arrhythmias
* No NYHA Class > II CHF
* No uncontrollable supraventricular arrhythmias
* No history of a ventricular arrhythmia
* No other clinical signs of severe cardiac dysfunction
* Normal Transthoracic Echocardiogram (TTE) is required for patients who have history of EKG abnormalities, CHF, coronary artery disease or other cardiac disease, or have history of having received adriamycin or doxorubicin
* No patients with a left ventricular ejection fraction (LVEF) of less than 50%

Pulmonary

• Normal clinical assessment of pulmonary function

Other

* Negative serum pregnancy test if female and of childbearing potential
* Women who are not pregnant or nursing
* Subjects, both females and males, with reproductive potential must agree to use effective contraceptive measures for the duration of the study
* No known autoimmune disease other than corrected hypothyroidism
* No known prior organ allograft or allogeneic transplantation
* Not HIV positive
* No active systemic infection requiring parenteral antibiotic therapy
* No ongoing systemic steroid therapy required
* No history or evidence of uncontrollable CNS disease
* No psychiatric illness/social situation
* No other illness that in the opinion of the investigator would exclude the subject from participating in the study
* Must provide informed consent and HIPAA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of California Davis, Sacramento, California
  - UF Health Center at Orlando Health, Orlando, Florida
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - UPMC Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only Phase 1B was enrolled, no subjects were enrolled in Phase 2.
Period: Overall Study
Arm/Group | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine
Started | 9 | 3
Completed | 2 | 2
Not Completed | 7 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Study Terminated by Investigator | 2 | 0
Not completed — Disease Progression | 2 | 0
Not completed — PI and subject decided to terminate treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (11.36) | 71.0 (4.36) | 65.1 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Patients with Bacillus Calmette-Guerin (BCG) Failure Non-Muscle Invasive Bladder Cancer [Count of Participants; unit: Participants] | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile
Description: Confirmation of the safety and tolerability (dose limiting toxicity count) of ALT-801 combined with gemcitabine.
Time Frame: 12 weeks
Measure: Number; unit: Number of DLTs
Arm/Group | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine
Number analyzed (Participants) | 9 | 3
Number of DLTs | 2 | 1

2. Primary Outcome: Disease Response Rate
Description: The response rate was calculated as the ratio of the number of patients who demonstrated a complete response (by RECIST v1.1) divided by the number of patients evaluable for response. A complete response was defined as having negative bladder biopsy results.
Time Frame: From start of study treatment to up to 13 weeks
Population: The population only included patients evaluable for response. 2 participants had no disease response information provided.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine
Number analyzed (Participants) | 7 | 3
percentage of participants | 43 [9.9 to 81.6] | 67 [9.4 to 99.2]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the date of first complete response (by RECIST v1.1) to the date of disease progression (by RECIST v1.1) or death (from any cause), whichever occured first. A complete response was defined as having negative bladder biopsy results. Disease progression by RECIST v1.1 is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression.
Time Frame: From confirmed complete response to up to 3 years
Population: Subjects with complete response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine
Number analyzed (Participants) | 3 | 2
Months | NA [5.2 to NA] — NA = not calculable due to small number of complete responders | 2.1 [1.2 to NA] — NA = not calculable due to small number of complete responders

4. Secondary Outcome: Progression-free Survival
Description: The progression-free survival was defined as the time from the start of study treatment to first documentation of objective tumor progression or disease recurrence (by RECIST v1.1). Disease progression by RECIST v1.1 is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression.
Time Frame: From start of study treatment to up to 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine
Number analyzed (Participants) | 7 | 3
Months | 3.4 [1.7 to NA] — not calculable due to small sample size and small number of subjects with events | 2.9 [2.7 to NA] — not calculable due to small sample size and small number of subjects with events

5. Secondary Outcome: Event-free Survival
Description: The event-free survival was defined as the time from the start of study treatment to first documentation of objective tumor progression (by RECIST v1.1), disease recurrence, bladder resection or irradiation, other anti-bladder cancer therapy, or to death due to any cause, which ever came first. Disease progression by RECIST v1.1 is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression.
Time Frame: From start of study treatment to up to 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine
Number analyzed (Participants) | 7 | 3
Months | 3.4 [1.7 to NA] — not calculable due to small sample size and small number of subjects with events | 2.9 [2.7 to NA] — not calculable due to small sample size and small number of subjects with events

6. Secondary Outcome: Overall Survival
Description: OS was defined as the time from start of study treatment to death resulting from any cause.
Time Frame: From start of study treatment to up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine
Number analyzed (Participants) | 9 | 3
Months | NA [7.5 to NA] — not calculable due to small sample size and small number of subjects with events | NA [21.2 to NA] — not calculable due to small sample size and small number of subjects with events

ADVERSE EVENTS:
Time Frame: For AEs and SAEs: 30 days past treatment completion, up to 16 weeks. For all cause mortality: from start of treatment up to approximately 3 years.
Arm/Group | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine
All-Cause Mortality (participants affected / at risk) | 2/9 | 1/3
Serious Adverse Events (participants affected / at risk) | 3/9 | 1/3
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine (N=9) | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine (N=3)
Skin Infection (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Anaphylaxis (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.06 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine (N=9) | 0.08 mg/kg ALT-801 With 1000 mg/m^2 Gemcitabine (N=3)
Chills (General disorders) | 7 | 2
Fatigue (General disorders) | 6 | 2
Edema limbs (General disorders) | 4 | 2
Fever (General disorders) | 3 | 2
Dry skin (General disorders) | 1 | 0
Flu like symptoms (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
General disorders and administration site conditions-other, feeling cold (General disorders) | 1 | 0
General disorders and administration site conditions-other, upper lip swelling (General disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Rash mucula-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash on thigh, back and buttocks (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders-other, gritty, sandpaper feeling between fingers (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders-other, hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
Alannine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Asparte aminotransferase increased (Investigations) | 1 | 0
Weight gain (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Nervous system disorders, other-numbness (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Tremors (Nervous system disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 2
Hot flashes (Vascular disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (non specific) (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Difficulty swallowing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Acute kidney disease (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Renal and urinary disorders, other-pyuria (Renal and urinary disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Eye disorders-other, visual disturbances (Eye disorders) | 1 | 0
Elevated alanine aminotransferase (Hepatobiliary disorders) | 1 | 0
Elevated Aspartate aminotransferase (Hepatobiliary disorders) | 1 | 0
Increased bilirubin (Hepatobiliary disorders) | 1 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Gemcitabine dosing was added in version 3 of the study protocol. 2 subjects were enrolled in protocol versions 1 and 2, which is why these subjects did not receive gemcitabine.

The study was terminated early due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT01625260/Prot_SAP_000.pdf